CLINICAL TRIAL: NCT06933069
Title: A Multicenter, Open-label Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Preliminary Anti-tumor Activity of CMAB017 in Advanced Malignant Solid Tumors
Brief Title: Safety and Tolerability of CMAB017 In Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMAB017-001
Record Dates: First submitted 2025-04-01; First posted 2025-04-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Solid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMAB017 (Experimental): CMAB017 100 mg intravenous (IV) solution for Injection every 3 weeks (Q3W) or every 2 weeks (Q2W)
  Interventions: Drug: CMAB017

INTERVENTIONS:
Drug: CMAB017 — CMAB017 was administered at a preset dose, and body weight was measured before each study dose; if body weight changed ≥10% from baseline, the dose should be recalculated. Administration was by intravenous infusion: for doses ≤1000 mg, intravenous infusion lasted 60±5 min; for doses >1000 mg, intravenous infusion lasted 90±5 min.

SUMMARY:
This is a multicenter, open-lable phase Ia clinical study to evaluate the safety, tolerability, pharmacokinetic profile and preliminary antitumor activity of CMAB017 in advanced malignant solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-lable, phase Ia study of CMAB017 which is planned to enroll about 55 patients with advanced solid tumors. The study is divided into the core period and the extension period.The core period involves the first four administrations of the drug, divided into two cohorts: the Q3W cohort (administering once every three weeks) and the Q2W cohort (administering once every two weeks). The pharmacokinetic profile and immunogenicity after completing dose escalation and observation for a total of four administrations are to be evaluated. In the extension period, for those subjects with therapeutic effects and tolerable side effects, the drug administration is to be prolonged. Further observations are to be made on the long-term safety, pharmacokinetic characteristics, immunogenicity, and anti-tumor effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. fully understand and agree to sign the Informed Consent Form (ICF);
2. histologically or cytologically confirmed, inoperable, locally advanced, recurrent or metastatic malignant solid tumors, including but not limited to head and neck squamous carcinoma, RAS wild-type colorectal cancer, esophageal squamous carcinoma, etc., for which the patient has failed standard treatment, does not have standard treatment, or refuses standard treatment;
3. age 18~75 years old, gender is not limited;
4. Eastern Cooperative Oncology Group (ECOG) score ≤1;
5. expected survival ≥ 3 months;
6. presence of at least one evaluable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 (bone-only metastases or central nervous system-only metastases will not be accepted as evaluable lesions); starting from 6 mg/kg Q3W, 4 mg/kg Q2W after the start of the dose group, presence of at least one measurable lesion; and dose groups, at least one measurable lesion is present (bone-only metastases or CNS-only metastases will not be accepted as measurable lesions);
7. females of childbearing potential must be non-lactating and have a negative serum pregnancy test within 1 week prior to the first infusion and agree to use effective contraception from the time of signing the ICF until 6 months after the last infusion; male subjects must agree to use effective contraception from the time of signing the ICF until 6 months after the last infusion;
8. Blood routine and liver and kidney functions during the screening period meet the following conditions:

   * Blood routine: neutrophils ≥1.5×109/L; platelets ≥75×109/L; hemoglobin ≥90 g/L;

     * Liver function: alanine aminotransferase and aspartate aminotransferase ≤3×ULN (both should be ≤5×ULN for those with tumor liver metastasis); total bilirubin ≤1.5×ULN; ③ Coagulation function: activated partial thromboplastin time (APTT) ≤1.5×ULN; international normalized ratio (INR) ≤1.5×ULN (for patients not receiving anticoagulation therapy; APTT or INR of subjects receiving anticoagulation therapy should be within the expected therapeutic range of anticoagulant drugs); ④ Renal function: blood creatinine ≤ 1.5 x ULN; if creatinine > 1.5 x ULN, creatinine clearance (Ccr) > 50mL/min is required (calculated according to the Cockcroft-Gault formula).

Exclusion Criteria:

1. With known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may be enrolled in the study provided that they have been clinically stable for at least 2 weeks, have no evidence of new or expanding brain metastases, and have discontinued steroids within 2 weeks prior to the infusion of the trial drug. Stability of brain metastases should be determined prior to the first dose of the trial drug infusion. Patients with asymptomatic brain metastases (i.e., no neurologic symptoms, no need for medication, and no lesion with a longest diameter >1.5 cm) may be enrolled, but will be required to undergo periodic imaging;
2. subjects with grade ≥2 corneal abnormalities present at screening;
3. adverse effects of prior antineoplastic therapy that have not recovered to a CTCAE 5.0 grade rating of ≤ grade 1 or to the level specified in the entry criteria (except for toxicities judged by the investigator to be of no safety risk, e.g., alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stabilized by hormone replacement therapy)
4. other malignancies within the previous 5 years, usually with the exception of the following: a. any other aggressive malignancy (for which the subject has had adequate treatment) for which disease-free status has persisted for >3 years and which, in the investigator's assessment, would not interfere with the assessment of oncologic efficacy; and b. cured basal cell or squamous cell skin cancers, superficial bladder cancers, and locally curable cancers such as prostate, cervical, or breast cancer in situ;
5. a history of immunodeficiency, including a positive HIV antibody test, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation
6. interstitial lung disease that is symptomatic or may interfere with pulmonary toxicity monitoring associated with the test drug;
7. a history of serious cardiovascular or cerebrovascular disease, including, but not limited to: severe cardiac rhythm or conduction block, such as ventricular arrhythmia requiring clinical intervention, degree III atrioventricular block, etc.; QTc intervals > 480 ms on 12/15 lead ECG at rest; acute coronary syndrome, congestive heart failure, aortic dissection, stroke within 6 months prior to the first infusion or other grade 3 or higher cardiovascular events; NYHA cardiac function classification ≥ grade II or LVEF <50%; clinically uncontrollable hypertension;
8. any of the following within 4 weeks prior to the first trial drug infusion:

   * Has had major surgery (defined as surgery requiring general anesthesia).
   * has participated in a clinical trial and received investigational treatment or used an investigational device.
   * Undergoing or planning other antineoplastic therapy outside of this study protocol (certain specific antineoplastic agents may be excluded from the 4 weeks prior to drug infusion, e.g., oral fluorouracil ≥ 2 weeks; mitomycin C, nitrosoureas ≥ 6 weeks; and small molecule targeted therapy ≥ 2 weeks);
9. any of the following within 2 weeks prior to the first trial drug infusion:

   * Having had localized palliative radiotherapy.
   * Received herbal/proprietary Chinese medicines that are clearly indicated for the treatment of oncological indications.
   * Has had minor surgery (other than major surgery, but diagnostic procedures such as incision and/or needle core biopsy are not considered minor surgery).
   * Received blood transfusion, erythropoietin, granulocyte colony-stimulating factor or granulocyte-macrophage colony-stimulating factor therapy;
10. known intolerance to anti-EGFR monoclonal antibodies resulting in discontinuation due to rash, gastrointestinal toxicity, or other Grade 3 or 4 toxicity;
11. Hepatitis B or C virologic testing at screening meets any of the following:

    * HBsAg positive and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV-DNA) titer test ≥1000 copies/mL or ≥200 IU/mL;
    * Positive antibody to HCV;
12. known severe allergic reaction to any component of the test drug or multiple drugs;
13. third interstitial fluid that, in the opinion of the investigator, is clinically uncontrollable;
14. any other serious or uncontrollable medical condition, active infection currently requiring intravenous anti-infective therapy, abnormal physical examination, abnormal laboratory tests, abnormal mental status, or psychiatric illness that, in the opinion of the Investigator, results in increased risk to the subject or otherwise affects the evaluation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities，DLT | Up to 12 weeks
Maximal Tolerated Dose，MTD | Up to 12 weeks

SECONDARY OUTCOMES:
Safety: The severity and incidence of other adverse events (AE) outside DLT | Date of the first dosing of study drug to 28 days post last dose of study drug.
Peak blood Concentration (Cmax) | Day 1 to Day 15
Trough blood Concentration (Cmin) | Day 1 to Day 15
Steady-state area under the plasma concentration versus time curve (AUC0-τ) | Day 1 to Day 15
Half life (t1/2) | Day 1 to Day 15
Time to reach maximum concentration (Tmax) | Day 1 to Day 15
Clearance (CL） | Day 1 to Day 15
Steady-state apparent volume of distribution (Vss) | Day 1 to Day 15
Immunogenicity: The occurrence rate of ADA and neutralizing antibody (Nab) | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No